CLINICAL TRIAL: NCT01186939
Title: AZA PH GL 2003 CL 001 - Extension A Multicenter, Randomized, Open-label, Parallel-group, Phase 3 Trial of Subcutaneous Azacitidine Plus Best Supportive Care Versus Conventional Care Regimens Plus Best Supportive Care for the Treatment of Myelodysplastic Syndromes (MDS)
Brief Title: An Extension to Study AZA PH GL 2003 CL 001 Allowing for Continuation of Azacitidine Treatment in Patients With Myelodysplastic Syndromes (MDS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZA PH GL 2003 CL001 E
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Results first posted 2010-09-21 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azacitidine (Experimental): Azacitidine (study drug) plus best supportive care.
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — Azacitidine was injected subcutaneously (SC) for 7 days. The 7-day dosing was repeated every 28 days with dose adjustments allowed. The initial dose during the primary study was 75mg/m^2/day.
  Other Names: AZA

SUMMARY:
At the conclusion of study AZA PH GL 2003 CL 001 (NCT00071799), eligible participants could be enrolled in an optional extension phase in order to continue treatment with azacitidine until it became commercially available; the continued treatment was for ethical and safety reasons only and not to provide additional efficacy data.

DETAILED DESCRIPTION:
At the conclusion of study AZA PH GL 2003 CL 001 (NCT00071799), eligible participants could be enrolled in an optional extension phase in order to continue treatment with azacitidine until it became commercially available; the continued treatment was for ethical and safety reasons only and not to provide additional efficacy data.

During the extension phase, participants were treated based on 28-day cycles and monitored for hematologic, nonhematologic, and renal toxicities. Recommended monitoring procedures included complete blood count with differential and platelets at least once each cycle prior to dosing and as needed, bone marrow biopsy and aspirate as clinically indicated, and additional tests or more frequent monitoring at the investigator's discretion based on the patient's clinical status. The azacitidine dose could be modified for toxicities. Laboratory data were not collected during the extension phase.

ELIGIBILITY:
Inclusion Criteria:

* Participants were considered eligible if they had been randomized to azacitidine treatment in the primary study and were receiving azacitidine at the time of study closure, had completed 12 months of treatment and observation in the primary study, and had signed the informed consent document for the extension phase of the study.
* See study: AZA PH GL 2003 CL 001 for a list of inclusion criteria for the primary study.

Exclusion Criteria:

* None specific to the extension phase of the study
* See study: AZA PH GL 2003 CL 001 for a list of exclusion criteria for the primary study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2009-09-01 (Actual); Study Completion 2009-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- Australia (4):
  - East Melbourne, Victoria
  - Herston
  - Perth
  - Woolloongabba
- Plovdiv, Bulgaria
- Aulnay-sous-Bois, France
- Germany (4):
  - Berlin
  - Düsseldorf
  - Essen
  - Kiel
- Greece (2):
  - Heraklio, Crete
  - Haidari
- Budapest, Hungary
- Italy (4):
  - Bologna
  - Florence
  - Genova
  - Rome
- Nijmegen, Netherlands
- Lodz, Poland
- Spain (2):
  - Avda Campanar
  - León
- London, United Kingdom

REFERENCES:
- [Background] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Finelli C, Giagounidis A, Schoch R, Gattermann N, Sanz G, List A, Gore SD, Seymour JF, Bennett JM, Byrd J, Backstrom J, Zimmerman L, McKenzie D, Beach C, Silverman LR; International Vidaza High-Risk MDS Survival Study Group. Efficacy of azacitidine compared with that of conventional care regimens in the treatment of higher-risk myelodysplastic syndromes: a randomised, open-label, phase III study. Lancet Oncol. 2009 Mar;10(3):223-32. doi: 10.1016/S1470-2045(09)70003-8. Epub 2009 Feb 21. PMID 19230772
- [Background] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Gattermann N, Germing U, Sanz G, List AF, Gore S, Seymour JF, Dombret H, Backstrom J, Zimmerman L, McKenzie D, Beach CL, Silverman LR. Azacitidine prolongs overall survival compared with conventional care regimens in elderly patients with low bone marrow blast count acute myeloid leukemia. J Clin Oncol. 2010 Feb 1;28(4):562-9. doi: 10.1200/JCO.2009.23.8329. Epub 2009 Dec 21. PMID 20026804
- [Background] Gore SD, Fenaux P, Santini V, Bennett JM, Silverman LR, Seymour JF, Hellstrom-Lindberg E, Swern AS, Beach CL, List AF. A multivariate analysis of the relationship between response and survival among patients with higher-risk myelodysplastic syndromes treated within azacitidine or conventional care regimens in the randomized AZA-001 trial. Haematologica. 2013 Jul;98(7):1067-72. doi: 10.3324/haematol.2012.074831. Epub 2013 Apr 12. PMID 23585522
- [Background] Savona MR, Kolibaba K, Conkling P, Kingsley EC, Becerra C, Morris JC, Rifkin RM, Laille E, Kellerman A, Ukrainskyj SM, Dong Q, Skikne BS. Extended dosing with CC-486 (oral azacitidine) in patients with myeloid malignancies. Am J Hematol. 2018 Oct;93(10):1199-1206. doi: 10.1002/ajh.25216. Epub 2018 Sep 3. PMID 30016552
- [Background] Seymour JF, Fenaux P, Silverman LR, Mufti GJ, Hellstrom-Lindberg E, Santini V, List AF, Gore SD, Backstrom J, McKenzie D, Beach CL. Effects of azacitidine compared with conventional care regimens in elderly (>/= 75 years) patients with higher-risk myelodysplastic syndromes. Crit Rev Oncol Hematol. 2010 Dec;76(3):218-27. doi: 10.1016/j.critrevonc.2010.04.005. Epub 2010 May 6. PMID 20451404
- [Background] Garcia-Manero G, Scott BL, Cogle CR, Boyd TE, Kambhampati S, Hetzer J, Dong Q, Kumar K, Ukrainskyj SM, Beach CL, Skikne BS. CC-486 (oral azacitidine) in patients with myelodysplastic syndromes with pretreatment thrombocytopenia. Leuk Res. 2018 Sep;72:79-85. doi: 10.1016/j.leukres.2018.08.001. Epub 2018 Aug 3. PMID 30114559
- [Background] Ma X, Steensma DP, Scott BL, Kiselev P, Sugrue MM, Swern AS. Selection of patients with myelodysplastic syndromes from a large electronic medical records database and a study of the use of disease-modifying therapy in the United States. BMJ Open. 2018 Jul 23;8(7):e019955. doi: 10.1136/bmjopen-2017-019955. PMID 30037860
- [Background] de Lima M, Oran B, Champlin RE, Papadopoulos EB, Giralt SA, Scott BL, William BM, Hetzer J, Laille E, Hubbell B, Skikne BS, Craddock C. CC-486 Maintenance after Stem Cell Transplantation in Patients with Acute Myeloid Leukemia or Myelodysplastic Syndromes. Biol Blood Marrow Transplant. 2018 Oct;24(10):2017-2024. doi: 10.1016/j.bbmt.2018.06.016. Epub 2018 Jun 20. PMID 29933073
- [Background] Wehmeyer J, Zaiss M, Losem C, Schmitz S, Niemeier B, Harde J, Hannig CV, Harich HD, Muller J, Klausmann M, Tessen HW, Potthoff K. Impact of performance status and transfusion dependency on outcome of patients with myelodysplastic syndrome, acute myeloid leukemia and chronic myelomonocytic leukemia treated with azacitidine (PIAZA study). Eur J Haematol. 2018 Dec;101(6):766-773. doi: 10.1111/ejh.13160. Epub 2018 Oct 25. PMID 30091166
- [Background] Platzbecker U, Middeke JM, Sockel K, Herbst R, Wolf D, Baldus CD, Oelschlagel U, Mutherig A, Fransecky L, Noppeney R, Bug G, Gotze KS, Kramer A, Bochtler T, Stelljes M, Groth C, Schubert A, Mende M, Stolzel F, Borkmann C, Kubasch AS, von Bonin M, Serve H, Hanel M, Duhrsen U, Schetelig J, Rollig C, Kramer M, Ehninger G, Bornhauser M, Thiede C. Measurable residual disease-guided treatment with azacitidine to prevent haematological relapse in patients with myelodysplastic syndrome and acute myeloid leukaemia (RELAZA2): an open-label, multicentre, phase 2 trial. Lancet Oncol. 2018 Dec;19(12):1668-1679. doi: 10.1016/S1470-2045(18)30580-1. Epub 2018 Nov 12. PMID 30442503
- [Background] Boutault R, Peterlin P, Boubaya M, Sockel K, Chevallier P, Garnier A, Guillaume T, Le Bourgeois A, Debord C, Godon C, Le Bris Y, Theisen O, Kroschinsky F, Moreau P, Bene MC, Platzbecker U, Eveillard M. A novel complete blood count-based score to screen for myelodysplastic syndrome in cytopenic patients. Br J Haematol. 2018 Dec;183(5):736-746. doi: 10.1111/bjh.15626. Epub 2018 Nov 8. PMID 30406952
- [Background] Wenk C, Garz AK, Grath S, Huberle C, Witham D, Weickert M, Malinverni R, Niggemeyer J, Kyncl M, Hecker J, Pagel C, Mulholland CB, Muller-Thomas C, Leonhardt H, Bassermann F, Oostendorp RAJ, Metzeler KH, Buschbeck M, Gotze KS. Direct modulation of the bone marrow mesenchymal stromal cell compartment by azacitidine enhances healthy hematopoiesis. Blood Adv. 2018 Dec 11;2(23):3447-3461. doi: 10.1182/bloodadvances.2018022053. PMID 30518537
- [Background] Zeidan AM, Klink AJ, McGuire M, Feinberg B. Treatment sequence of lenalidomide and hypomethylating agents and the impact on clinical outcomes for patients with myelodysplastic syndromes. Leuk Lymphoma. 2019 Aug;60(8):2050-2055. doi: 10.1080/10428194.2018.1551538. Epub 2019 Jan 14. PMID 30636526
- [Background] Leung KK, Nguyen A, Shi T, Tang L, Ni X, Escoubet L, MacBeth KJ, DiMartino J, Wells JA. Multiomics of azacitidine-treated AML cells reveals variable and convergent targets that remodel the cell-surface proteome. Proc Natl Acad Sci U S A. 2019 Jan 8;116(2):695-700. doi: 10.1073/pnas.1813666116. Epub 2018 Dec 24. PMID 30584089
- [Background] Craddock C, Slade D, De Santo C, Wheat R, Ferguson P, Hodgkinson A, Brock K, Cavenagh J, Ingram W, Dennis M, Malladi R, Siddique S, Mussai F, Yap C. Combination Lenalidomide and Azacitidine: A Novel Salvage Therapy in Patients Who Relapse After Allogeneic Stem-Cell Transplantation for Acute Myeloid Leukemia. J Clin Oncol. 2019 Mar 1;37(7):580-588. doi: 10.1200/JCO.18.00889. Epub 2019 Jan 17. PMID 30653424
- [Result] Silverman LR, Fenaux P, Mufti GJ, Santini V, Hellstrom-Lindberg E, Gattermann N, Sanz G, List AF, Gore SD, Seymour JF. Continued azacitidine therapy beyond time of first response improves quality of response in patients with higher-risk myelodysplastic syndromes. Cancer. 2011 Jun 15;117(12):2697-702. doi: 10.1002/cncr.25774. Epub 2011 Jan 10. PMID 21656747
- See also: Study record for primary study — http://www.clinicaltrials.gov/ct2/results?term=NCT00071799

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were eligible for the extension study of AZA PH GL 2003 CL 001 if they had been randomized to azacitidine treatment in the primary study and receiving azacitidine at the time of study closure, completed 12 months of treatment and observation in the primary study, and signed the informed consent document for the extension study.
Groups:
- Azacitidine: Azacitidine (study drug) plus best supportive care. Azacitidine was injected subcutaneously (SC) for 7 days. The 7-day dosing was repeated every 28 days with dose adjustments allowed. The initial dose during the primary study was 75mg/m^2/day.
Period: Overall Study
Arm/Group | Azacitidine
Started | 40
Completed | 0
Not Completed | 40
Not completed — Death | 7
Not completed — Withdrawal by Subject | 2
Not completed — No longer receiving clinical benefit | 17
Not completed — Program closed | 5
Not completed — Sponsor decision | 4
Not completed — Started additional treatment | 1
Not completed — NCI CTC Grade 3 or 4 toxicity | 1
Not completed — Myocardial infarction | 1
Not completed — Bone marrow transplant | 1
Not completed — Transformation to AML | 1

BASELINE CHARACTERISTICS:
Arm/Group | Azacitidine
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (8.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 32
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 40
French-American-British (FAB) Classification [Number; unit: participants] — FAB classifications were determined by the Independent Review Committee
  participants
    Refractory anemia with excess blasts (RAEB) | 27
    RAEB in transformation | 10
    Modified chronic myelomonocytic leukemia | 1
    Acute myeloid leukemia | 1
    Myeloproliferative disease | 1
World Health Organization (WHO) Classification [Number; unit: participants] — WHO classifications were determined by the Independent Review Committee.
  participants
    Refractory anemia with excess blasts - 1 | 5
    Refractory anemia with excess blasts - 2 | 22
    Chronic myelomonocytic leukemia - 1 (CMMoL-1) | 0
    Chronic myelomonocytic leukemia - 2 (CMMoL-2) | 2
    Acute myeloid leukemia | 11
International Prognostic Scoring System (IPSS) [Number; unit: participants] — The international prognostic scoring system (IPSS) is a standard for risk assessment in primary myelodysplastic syndromes (MDS) that categorizes prognoses taking into account cytogenetics, cytopenias, blasts and blood counts. The scale is 0-3.5 at .5 increments. Scores of 2.5-3.5 represent high risk which corresponds to poorer prognosis. The assessment was performed by the Independent Review Committee.
  participants
    Intermediate risk level 1 (0.5-1.0) | 1
    Intermediate risk level 2 (1.5-2.0) | 21
    High risk (2.5-3.5) | 14
    Not applicable | 2
    Indeterminate | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Different Categories of Treatment Emergent Adverse Events for the Extension Period
Description: Participant counts for a variety of subsets of treatment emergent adverse events (TEAEs)during the extension study period (43-68 months). Subsets include participants counts for serious TEAEs, serious TEAEs that the investigator evaluated as releated to treatment, TEAEs leading to discontinuation of therapy, or a dose reduction, or a dose interruption.
Time Frame: 43- 68 months
Population: Safety population includes all 40 participants in the extension study.
Measure: Number; unit: participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 40
participants
  Participants with >=1 treatment emergent AE (TEAE) | 39
  Participants with >=1 treatment related TEAE | 27
  Participants with >=1 serious TEAE | 20
  Participants with >=1 serious trtment related TEAE | 5
  Participants w TEAE leading to discontinued treat | 15
  Participants w TEAE leading to dose reduction | 4
  Participants w TEAE leading to dose interruption | 15

ADVERSE EVENTS:
Time Frame: Extension study covering 43- 68 months
Description: Includes adverse events that started up to 42 days after the date of last dose of azacitidine in the extension study. Also any adverse event that started outside the treatment-emergent periods and assessed as related to study drug is considered treatment emergent.
Arm/Group | Azacitidine
Serious Adverse Events (participants affected / at risk) | 20/40
Other Adverse Events (participants affected / at risk) | 36/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine (N=40)
Anaemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 1
Pyrexia (General disorders) | 1
Injection site infection (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Perianal abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
White blood cell count increase (Investigations) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Mental disorder due to a general medical condition (Psychiatric disorders) | 1
Renal artery stenosis (Renal and urinary disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Cardiovascular insufficiency (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine (N=40)
Anaemia (Blood and lymphatic system disorders) | 11
Leukopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 4
Fatigue (General disorders) | 6
Injection site erythema (General disorders) | 4
Injection site reaction (General disorders) | 8
Oedema peripheral (General disorders) | 5
Pyrexia (General disorders) | 7
Bronchitis (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Herpes virus infection (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 5
Oral herpes (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Depression (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Blood blister (Skin and subcutaneous tissue disorders) | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 2
Ecchmyosis (Skin and subcutaneous tissue disorders) | 3
Petechiae (Skin and subcutaneous tissue disorders) | 2
Haematoma (Vascular disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to publish and/or present study data provided that the investigator shall (i) furnish the sponsor a copy of any proposed publication or presentation generally thirty (30) days in advance of the submission, (ii) delete any confidential information of the sponsor, and (iii) delay submission for generally up to ninety (90) days to permit the preparation and filing of intellectual property applications or until sponsor gives its consent in a timely manner.